CLINICAL TRIAL: NCT06499012
Title: A Randomized, Double-blind Clinical Study of the Efficacy of Nutrilite All-plant Protein Booster to Improve Sarcopenia and Osteoarthritis in Middle-aged and Elderly People
Brief Title: The Efficacy of Nutrilite All-plant Protein Booster to Improve Sarcopenia and Osteoarthritis in Middle-aged and Elderly People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amway (China) R&D Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IS20220021RD
Record Dates: First submitted 2024-07-06; First posted 2024-07-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Osteoarthritis; Sarcopenia
Keywords: Amway Nutrilite; All-plant Protein Booster; SPPB; WOMAC; WHOQOL BREF; SF-36; CFQ 11; SFQ
MeSH Terms: conditions — Osteoarthritis; Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- All-plant Protein Booster Product Group (Active Comparator): Containing ingredients: Soy protein Isolate, Soybean peptide, wheat protein, pea protein, Pea peptide, Aloe Vera powder, Sweetener (Maltitol) Anti-caking (Silicon Dioxide) Thickener (guar gum, arabic gum)
  Interventions: Dietary Supplement: All-plant Protein Booster Product Group
- Placebo Group (Placebo Comparator): Containing ingredients: Aloe Vera powder, Sweetener (Maltitol) Anti-caking (Silicon Dioxide) Thickener (guar gum, arabic gum)
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: All-plant Protein Booster Product Group — Participants in this arm will take 2 spoons (15g) twice per day for 12 weeks
  Arms: All-plant Protein Booster Product Group
Dietary Supplement: Placebo Group — Participants in this arm will take 2 spoons (15g) twice per day for 12 weeks
  Arms: Placebo Group

SUMMARY:
The goal of this clinical trial is to learn whether Amway Nutrilite All-plant protein booster prototype product (test product) will improve sarcopenia (SA) and osteoarthritis (OA) in middle-aged and elderly people. It will also learn about the improvement of Quality of life (QoL) in them. The main questions it aims to answer are:

* Does the test product will improve the SA in terms of Short Physical Performance Battery (SPPB score) after 12 weeks' intervention?
* Does the test product will improve the OA in terms of Western Ontario and McMaster Universities Arthritis (WOMAC Index) after 12 weeks' intervention?

Researchers will compare Amway All-plant protein booster prototype product to a placebo (a look-alike substance that contains no similar active nutrient ingredients) to see if the test product works to improve SA and OA.

Participants will:

* Take the test product or a placebo 2 spoons (15g) twice per day for 12 weeks
* Visit the site on the baseline day and the 84th day (end day of 12 weeks) for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

* Be age 50 to 70 years, female and male
* Participants will be required to have mild to moderately OA & SA evaluated by Kellgren-Lawrence I-II and SARC-Cal, respectively
* Participants need to be competent i.e., able to understand what is to take place and able to provide a free decision on agreeing to the activity/taking part on the study on this
* Participants must be able to read and understand study instructions and any other relevant study documents
* Willing to following the lifestyle restrictions as detailed in the Information Sheet for study
* Will to give written informed consent

Exclusion Criteria:

* Have a fever currently, or for 24 hours before enrollment
* Currently participating in another clinical study
* Have taken other protein powder products and dietary supplements or medicines containing peptides or hyaluronic acid within the past 6 months (subject to product instructions)
* Individuals receiving medical treatment that, in the opinion of the Principal Investigator or Study Physician, may interfere with test results
* The participant is an employee of Amway or SPRIM Medical
* Subject who is in the treatment of gastrointestinal diseases
* Subject with abnormal liver function tests (alanine aminotransferase and aspartate aminotransferase), kidney function tests (blood urea nitrogen and creatinine), blood routine, urine routine, fecal occult blood test, or electrocardiogram.
* Subjects have any of the following medical history or have been clinically examined to have the following diseases that may affect the evaluation of the test effect: obvious gastrointestinal dysfunction, liver, kidney, endocrine, blood, respiratory and cardiovascular diseases

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2025-07-08 (Actual); Primary Completion 2025-10-02 (Actual); Study Completion 2025-10-02 (Actual)

PRIMARY OUTCOMES:
Change of SPPB Score from baseline | baseline day 0, week 12
  The SPPB (Short Physical Performance Battery) test is a group of measures that combines the results of the gait speed, chair stand and balance tests (Guralnik et al., 2000). lt has been used as a predictive tool for possible disability and can aid in the monitoring of function in older people. The scores range from 0 (worst performance) to 12 (best performance).
Change of WOMAC 3.1 index from baseline | baseline day 0, week 12
  The WOMAC (Western Ontario and McMaster Universities Arthritis) Index was created to assess pain, stiffness, and physical function in patients with hip and / or knee osteoarthritis (OA). The WOMAC 3.1 consists of 24 items divided into 3 subscales. The scores are summed for items in each subscale, with possible ranges as follows: pain=0-20, stiffness=0-8, physical function=0-68. A total WOMAC score is created by summing the items for all three subscales. (0-96), higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations.

SECONDARY OUTCOMES:
Change of bone density measured by DXA Bone Densitometer from baseline | baseline day 0, week 12
  Change of bone density measured by DXA Bone Densitometer from baseline to week 12
Improvement of Fat and Muscle Portions measured by Inbody S10 from baseline | baseline day 0, week 12
  Improvement of Fat and Muscle Portions measured by Inbody S10 from baseline to week 12
Improvement of Quality of Life by WHOQOL BREF | baseline day 0, week 12
  WHOQOL-BREF is a generic health related QoL measure consisting of 26 items divided into 6 sub-scales.
Improvement of Quality of Life by SF-36 | baseline day 0, week 12
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that comprises 36 questions that cover eight domains of health.
Improvement of Quality of Life by Chalder Fatigue Scale (CFQ 11) | baseline day 0, week 12
  Change of Chalder Fatigue Scale (CFQ 11), with range from 0 to 11 (the bigger the score, the more fatigue a person feels), from baseline to week 12. The Chalder fatigue scale (CFQ 11) is a questionnaire created by the research team of Trudie Chalder at King's College London to measure the severity of tiredness in fatiguing illnesses.
Change of SFQ from baseline | baseline day 0, week 12
  The change of frequency of sports activity by SFQ (Sports Frequency Questionnaire) from baseline to week 12

CONTACTS AND LOCATIONS:
Overall Officials: Zhenzhong Lu, MD, Principal Investigator — Jinhua Wenrong Hospital
Locations (1):
- Jinhua Wenrong Hospital, Jinhua, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No